CLINICAL TRIAL: NCT03721666
Title: Medical Dispatchers' Perception of Visual Information in Real Out-of-hospital Cardiac Arrest: A Qualitative Interview Study
Brief Title: Medical Dispatchers' Perception of Visual Information in Real Out-of-hospital Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Emergency Medical Services, Capital Region, Denmark (Other Government)
Collaborators: TrygFonden, Denmark (Industry); Danish Heart Foundation (Other)
Responsible Party: Principal Investigator, Gitte Linderoth, Principal Investigator, MD, Emergency Medical Services, Capital Region, Denmark
Other Study IDs: F-15035-02-GL
Record Dates: First submitted 2018-10-23; First posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2018-10

CONDITIONS: Out-Of-Hospital Cardiac Arrest
Keywords: Dispatcher-assisted cardiopulmonary resuscitation; Out-Of-Hospital Cardiac Arrest; Emergency Medical dispatcher
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: CCTV footage to the medical dispatcher in OHCA — The medical dispatchers' perception of bystanders' responses and dispatchers' reflections about the added value of visual information in out-of-hospital cardiac arrests (OHCA) situations.

SUMMARY:
Dispatcher-assisted cardiopulmonary resuscitation is a complex, nonvisual procedure that is challenging for the dispatcher. The aim was to explore the medical dispatchers' perception of bystanders' responses and dispatchers' reflections about the added value of visual information in out-of-hospital cardiac arrests (OHCA) situations.

DETAILED DESCRIPTION:
Ten individual interviews with medical dispatchers who had previously handled an emergency call concerning OHCA captured on closed-circuit television (CCTV) were conducted. First, the medical dispatcher listened to the emergency call and described their perception of the scenario. Afterward, the CCTV recording was shown to the dispatcher, who was then interviewed. The interviews were videotaped, and the audio files were transcribed verbatim. Thematic content analysis was conducted.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Medical dispatchers who had previously handled an emergency call concerning OHCA captured on closed-circuit television (CCTV)

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Emergency Medical dispatchers
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
The added value of visual information to the medical dispatcher in out-of-hospital cardiac arrests (OHCA) situations. | One hour interview with earch of the emergency medical dispathers
  We applied a qualitative research methodology using thematic analysis with an explorative and inductive approach. The first author followed Braun and Clarke's six-step analytical approach, which has the following steps: familiarising with data, generating initial codes, searching for themes, reviewing themes, defining and naming themes, and producing the report. Codes and themes were organised using Nvivo10 software (QSR International Pty Ltd, Australia). Analysis continued until saturation; that is, when information became redundant.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Oestergaard, Study Director — Copenhagen Academy for Medical Education and Simulation; Freddy K. Lippert, Study Chair — Emergency Medical Services, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
If other researchers want the themes and transcriptions it can be arranged.